CLINICAL TRIAL: NCT00826657
Title: Assessment of Functional Vitamin B12 Deficiency in Mexican Women
Brief Title: Vitamin B12 Supplementation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 200412519-3
Record Dates: First submitted 2009-01-16; First posted 2009-01-22 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Vitamin B12 Deficiency
Keywords: B12 deficiency; methylmalonic acid; homocystein; vitamin B12 supplementation intervention
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Vitamin B 12; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Receive placebo (sugar pill) during the intervention. Received a 1000 mg vitamin B12 injection at the end of the study.
  Interventions: Dietary Supplement: placebo
- Vitamin B12 (Active Comparator): Received 500 micrograms vitamin B12 per day during the study Received a 1000 mg vitamin B12 injection at the start of the study
  Interventions: Dietary Supplement: Vitamin B12

INTERVENTIONS:
Dietary Supplement: Vitamin B12 — 500 microgram daily supplement of vitamin B12 1000 mg injection vitamin B12 given at the start of the study
  Arms: Vitamin B12
Dietary Supplement: placebo — placebo given as a daily supplement 1000 mg injection of vitamin B12 given at the end of the study
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
We hope to learn the clinical and functional signs of sub-clinical vitamin B12 deficiency and its response to supplementation in non-anemic, non-pregnant, and non-lactating women in Rural Mexico. Vitamin B12 is important in hematopoiesis, neuro-cognitive functions and genetic integrity. However vitamin B12 is only found in animal source foods therefore a large segment of the population in developing countries and those practicing vegetarianism are at risk of deficiency of the vitamin. This information will help decide weather supplementation with vitamin B12 is necessary in such populations for public health reasons.

ELIGIBILITY:
Inclusion Criteria:

* Women age 20-59, apparently healthy, no severe B12 deficiency

Exclusion Criteria:

* pregnancy, lactation, anemia and disease states

Ages: 20 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2004-10; Primary Completion 2005-08 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
response to B12 supplementation in serum B12, Methylmalonic acid, homocystein, and holotranscobalamin concentrations | 0 and 3 mos

SECONDARY OUTCOMES:
DNA methylation change, and hematological response to B12 supplementation | 0 and 3 mos

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Autonoma de Queretaro, Querétaro, Mexico

REFERENCES:
- [Derived] Shahab-Ferdows S, Anaya-Loyola MA, Vergara-Castaneda H, Rosado JL, Keyes WR, Newman JW, Miller JW, Allen LH. Vitamin B-12 supplementation of rural Mexican women changes biochemical vitamin B-12 status indicators but does not affect hematology or a bone turnover marker. J Nutr. 2012 Oct;142(10):1881-7. doi: 10.3945/jn.112.165712. Epub 2012 Aug 22. PMID 22915298